CLINICAL TRIAL: NCT04015622
Title: A Randomized Phase II Trial Comparing Biomarker Directed Therapy Versus Clinician's Choice of Enzalutamide or Docetaxel in Patients With Advanced Prostate Cancer Post Abiraterone
Brief Title: PROstate Cancer TReatment Optimization Via Analysis of Circulating Tumour DNA
Acronym: PROTRACT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROTRACT
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: circulating tumor DNA; Enzalutamide; Docetaxel
MeSH Terms: interventions — enzalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Biomarker directed Therapy (BT) (Experimental): ctDNA fraction <2% receives enzalutamide, and ctDNA fraction ≥2% receives docetaxel until disease progression, then cross-over to the other therapy (e.g., enzalutamide to docetaxel, or docetaxel to enzalutamide).
  Interventions: Drug: Enzalutamide; Drug: Docetaxel
- B: Clinician's Choice (CC) (Active Comparator): Enzalutamide or docetaxel until disease progression, then cross-over to the other therapy (e.g., enzalutamide to docetaxel, or docetaxel to enzalutamide).
  Interventions: Drug: Enzalutamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide 160 mg PO OD
  Other Names: Xtandi
Drug: Docetaxel — Docetaxel 75 mg/m2 IV every 3 weeks
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to assess the strategy in treatment selection using ctDNA fraction as a predictive biomarker to direct treatment decision (ctDNA fraction <2% receives enzalutamide, and ctDNA fraction ≥2% receives docetaxel) versus clinician's choice of enzalutamide or docetaxel, in subjects with metastatic castration-resistant prostate cancer post abiraterone setting.

DETAILED DESCRIPTION:
This is a prospective, open-label, phase II trial with 1:1 randomization to either Arm A biomarker directed therapy (patients with ctDNA fraction <2% receive enzalutamide, and ctDNA fraction ≥2% receive docetaxel), versus Arm B clinician's choice of enzalutamide or docetaxel, in subjects with metastatic castration-resistant prostate cancer post abiraterone. At time of progression, patient will cross-over to the other therapy (e.g., enzalutamide to docetaxel, and docetaxel to enzalutamide).

ELIGIBILITY:
INCLUSION CRITERIA

Patients must meet ALL of the following criteria:

1. Willing and able to provide informed consent
2. Adult males ≥ 18 years age
3. History of histologically confirmed adenocarcinoma of the prostate without evidence of neuroendocrine or small cell differentiation. If histology is not available, patients must have metastatic disease typical of prostate cancer (i.e., involving bone or pelvic lymph nodes or para-aortic lymph nodes) AND a serum concentration of PSA that is rising and >20ng/mL at the time prostate cancer was diagnosed clinically
4. Consent to analysis of archival tissue collected at diagnosis is mandatory
5. Prior surgical orchiectomy or if on LHRH agonist/antagonist then testosterone < 1.7 nmol/L at screening visit (patients must maintain LHRH agonist/antagonist therapy for duration of study treatment if not surgically castrated)
6. Evidence of metastatic disease on bone scan or CT scan
7. Evidence of biochemical or imaging progression in the setting of surgical or medical castration while on abiraterone. Progressive disease for study entry is defined by one of the following three criteria as per PCWG317:

   1. PSA progression: minimum of two rising PSA values from a baseline measurement of one week interval. Minimum PSA at screening visit is 1.0 ng/mL
   2. Soft tissue or visceral disease progression: an increase ≥20% in the sum of the diameter (short axis for nodal lesions and long axis for non-nodal lesions) from the smallest sum of the diameter since treatment started, or appearance of any new lesions (see Appendix B for definition of measurable disease as per RECIST 1.1 criteria).
   3. Bone progression: ≥ 2 new lesions on bone scan confirmed on subsequent bone scan at least 8 weeks apart (2+2 rule as per PCWG317)
8. ECOG performance status 0-2 (see Appendix C)
9. Prior treatment with abiraterone, in either castration-sensitive or castration-resistant setting.
10. Eligible for treatment with either enzalutamide or docetaxel as per standard of care guidelines
11. Adequate organ function defined as:

    1. Absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L and hemoglobin ≥ 90 g/L
    2. Creatinine clearance ≥ 30 ml/min (calculated by Cockcroft-Gault formula, see Appendix D)
    3. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome (direct bilirubin ≤ 1.5 x ULN)
    4. Alanine aminotransferase (ALT) ≤ 5 x ULN
12. Able to swallow study drug and comply with study requirements including provision of peripheral blood samples at specified time points for correlative studies
13. Recovery from all prior treatment-related toxicity to grade ≤ 2 (as per CTCAE 5.0)

EXCLUSION CRITERIA

Patients must NOT meet any of the following criteria:

1. Severe concurrent illness or co-morbid disease that would make the subject unsuitable for enrolment
2. Prior therapy with enzalutamide or other experimental anti-androgens (e.g. ARN-509, TOK-001)
3. Prior systemic chemotherapy with docetaxel or cabazitaxel (with the exception of: patients who were treated with docetaxel for castration sensitive disease and did not progress for at least 12 months after completion of docetaxel)
4. Active concurrent malignancy (with the exception of non-melanomatous skin cancer, or other solid tumours curatively treated with no evidence of disease for ≥3 years)
5. Wide-field radiotherapy or radioisotopes such as Strontium-89, or Radium-223 ≤ 28 days prior to starting study drug (limited-field palliative radiotherapy for up to 5 fractions prior to starting study drug is permitted)
6. Brain metastases or active epidural disease (treated epidural disease is permitted)
7. Contraindication to prednisone therapy including poorly controlled diabetes mellitus
8. History of seizure or seizure disorder, or history of any cerebrovascular event within 6 months of study entry.
9. Uncontrolled hypertension Grade ≥3 (i.e. systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg)
10. Gastrointestinal disorder affecting absorption
11. Major surgery within 4 weeks of starting study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 year
  PFS is defined as the time between the date of starting trial treatment to any of the following: clinical, PSA, radiographic progression, or death from any cause on first-line therapy

SECONDARY OUTCOMES:
Objective response | 1 year
  To determine the objective response as per RECIST 1.1 in patients treated with biomarker directed therapy vs. clinician's choice.
PSA response rate | 1 year
  PSA response rate is defined as the proportion of patients with a PSA decline (defined as a ≥30%, ≥50% and other declines in PSA from baseline) in mCRPC patients treated with biomarker directed therapy vs. clinician's choice.
Second progression free survival (PFS2) | 1 year
  PFS2 is defined as the time elapsed between the date of treatment commencement and the first documented evidence of any disease progression or death from any cause from cross-over second-line therapy.
Overall survival (OS) | 2 years
  OS is defined as time from treatment commencement to death of any cause of mCRPC patients treated with biomarker directed therapy vs. clinician's choice.
Clinical benefit rate (CBR) | 3 months
  CBR is defined as PSA or measurable radiological response of any duration or stable disease for ≥ 12 weeks (no symptomatic progression, PSA progression, or objective disease progression).
Correlation of specific ctDNA-based genomic alterations to treatment response | 1 year
  Among mCRPC patients receiving enzalutamide and docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (7):
- Canada (7):
  - BC Cancer - Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - BC Cancer - Centre for the North, Prince George, British Columbia
  - BC Cancer - Surrey Centre, Surrey, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, British Columbia
  - BC Cancer - Vancouver Centre, Vancouver, British Columbia
  - BC Cancer - Victoria Centre, Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario

REFERENCES:
- [Background] Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, Ozguroglu M, Ye D, Feyerabend S, Protheroe A, De Porre P, Kheoh T, Park YC, Todd MB, Chi KN; LATITUDE Investigators. Abiraterone plus Prednisone in Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2017 Jul 27;377(4):352-360. doi: 10.1056/NEJMoa1704174. Epub 2017 Jun 4. PMID 28578607
- [Background] James ND, de Bono JS, Spears MR, Clarke NW, Mason MD, Dearnaley DP, Ritchie AWS, Amos CL, Gilson C, Jones RJ, Matheson D, Millman R, Attard G, Chowdhury S, Cross WR, Gillessen S, Parker CC, Russell JM, Berthold DR, Brawley C, Adab F, Aung S, Birtle AJ, Bowen J, Brock S, Chakraborti P, Ferguson C, Gale J, Gray E, Hingorani M, Hoskin PJ, Lester JF, Malik ZI, McKinna F, McPhail N, Money-Kyrle J, O'Sullivan J, Parikh O, Protheroe A, Robinson A, Srihari NN, Thomas C, Wagstaff J, Wylie J, Zarkar A, Parmar MKB, Sydes MR; STAMPEDE Investigators. Abiraterone for Prostate Cancer Not Previously Treated with Hormone Therapy. N Engl J Med. 2017 Jul 27;377(4):338-351. doi: 10.1056/NEJMoa1702900. Epub 2017 Jun 3. PMID 28578639
- [Background] Attard G, Parker C, Eeles RA, Schroder F, Tomlins SA, Tannock I, Drake CG, de Bono JS. Prostate cancer. Lancet. 2016 Jan 2;387(10013):70-82. doi: 10.1016/S0140-6736(14)61947-4. Epub 2015 Jun 11. PMID 26074382
- [Background] Lorente D, Mateo J, Perez-Lopez R, de Bono JS, Attard G. Sequencing of agents in castration-resistant prostate cancer. Lancet Oncol. 2015 Jun;16(6):e279-92. doi: 10.1016/S1470-2045(15)70033-1. Epub 2015 May 27. PMID 26065613
- [Background] Wyatt AW, Gleave ME. Targeting the adaptive molecular landscape of castration-resistant prostate cancer. EMBO Mol Med. 2015 Jul;7(7):878-94. doi: 10.15252/emmm.201303701. PMID 25896606
- [Background] Robinson D, Van Allen EM, Wu YM, Schultz N, Lonigro RJ, Mosquera JM, Montgomery B, Taplin ME, Pritchard CC, Attard G, Beltran H, Abida W, Bradley RK, Vinson J, Cao X, Vats P, Kunju LP, Hussain M, Feng FY, Tomlins SA, Cooney KA, Smith DC, Brennan C, Siddiqui J, Mehra R, Chen Y, Rathkopf DE, Morris MJ, Solomon SB, Durack JC, Reuter VE, Gopalan A, Gao J, Loda M, Lis RT, Bowden M, Balk SP, Gaviola G, Sougnez C, Gupta M, Yu EY, Mostaghel EA, Cheng HH, Mulcahy H, True LD, Plymate SR, Dvinge H, Ferraldeschi R, Flohr P, Miranda S, Zafeiriou Z, Tunariu N, Mateo J, Perez-Lopez R, Demichelis F, Robinson BD, Schiffman M, Nanus DM, Tagawa ST, Sigaras A, Eng KW, Elemento O, Sboner A, Heath EI, Scher HI, Pienta KJ, Kantoff P, de Bono JS, Rubin MA, Nelson PS, Garraway LA, Sawyers CL, Chinnaiyan AM. Integrative clinical genomics of advanced prostate cancer. Cell. 2015 May 21;161(5):1215-1228. doi: 10.1016/j.cell.2015.05.001. PMID 26000489
- [Background] Chedgy EC, Annala M, Beja K, Warner EW, Gleave ME, Chi KN, Wyatt AW. Moving Toward Personalized Care: Liquid Biopsy Predicts Response to Cisplatin in an Unusual Case of BRCA2-Null Neuroendocrine Prostate Cancer. Clin Genitourin Cancer. 2016 Apr;14(2):e233-6. doi: 10.1016/j.clgc.2015.12.023. Epub 2015 Dec 24. No abstract available. PMID 26797585
- [Background] Lallous N, Volik SV, Awrey S, Leblanc E, Tse R, Murillo J, Singh K, Azad AA, Wyatt AW, LeBihan S, Chi KN, Gleave ME, Rennie PS, Collins CC, Cherkasov A. Functional analysis of androgen receptor mutations that confer anti-androgen resistance identified in circulating cell-free DNA from prostate cancer patients. Genome Biol. 2016 Jan 26;17:10. doi: 10.1186/s13059-015-0864-1. PMID 26813233
- [Background] Wyatt AW, Azad AA, Volik SV, Annala M, Beja K, McConeghy B, Haegert A, Warner EW, Mo F, Brahmbhatt S, Shukin R, Le Bihan S, Gleave ME, Nykter M, Collins CC, Chi KN. Genomic Alterations in Cell-Free DNA and Enzalutamide Resistance in Castration-Resistant Prostate Cancer. JAMA Oncol. 2016 Dec 1;2(12):1598-1606. doi: 10.1001/jamaoncol.2016.0494. PMID 27148695
- [Background] Azad AA, Volik SV, Wyatt AW, Haegert A, Le Bihan S, Bell RH, Anderson SA, McConeghy B, Shukin R, Bazov J, Youngren J, Paris P, Thomas G, Small EJ, Wang Y, Gleave ME, Collins CC, Chi KN. Androgen Receptor Gene Aberrations in Circulating Cell-Free DNA: Biomarkers of Therapeutic Resistance in Castration-Resistant Prostate Cancer. Clin Cancer Res. 2015 May 15;21(10):2315-24. doi: 10.1158/1078-0432.CCR-14-2666. Epub 2015 Feb 23. PMID 25712683
- [Background] Annala M, Struss WJ, Warner EW, Beja K, Vandekerkhove G, Wong A, Khalaf D, Seppala IL, So A, Lo G, Aggarwal R, Small EJ, Nykter M, Gleave ME, Chi KN, Wyatt AW. Treatment Outcomes and Tumor Loss of Heterozygosity in Germline DNA Repair-deficient Prostate Cancer. Eur Urol. 2017 Jul;72(1):34-42. doi: 10.1016/j.eururo.2017.02.023. Epub 2017 Mar 1. PMID 28259476
- [Background] Quigley D, Alumkal JJ, Wyatt AW, Kothari V, Foye A, Lloyd P, Aggarwal R, Kim W, Lu E, Schwartzman J, Beja K, Annala M, Das R, Diolaiti M, Pritchard C, Thomas G, Tomlins S, Knudsen K, Lord CJ, Ryan C, Youngren J, Beer TM, Ashworth A, Small EJ, Feng FY. Analysis of Circulating Cell-Free DNA Identifies Multiclonal Heterogeneity of BRCA2 Reversion Mutations Associated with Resistance to PARP Inhibitors. Cancer Discov. 2017 Sep;7(9):999-1005. doi: 10.1158/2159-8290.CD-17-0146. Epub 2017 Apr 27. PMID 28450426
- [Background] Wyatt AW, Annala M, Aggarwal R, Beja K, Feng F, Youngren J, Foye A, Lloyd P, Nykter M, Beer TM, Alumkal JJ, Thomas GV, Reiter RE, Rettig MB, Evans CP, Gao AC, Chi KN, Small EJ, Gleave ME. Concordance of Circulating Tumor DNA and Matched Metastatic Tissue Biopsy in Prostate Cancer. J Natl Cancer Inst. 2017 Dec 1;109(12):djx118. doi: 10.1093/jnci/djx118. PMID 29206995
- [Background] Annala M, Vandekerkhove G, Khalaf D, Taavitsainen S, Beja K, Warner EW, Sunderland K, Kollmannsberger C, Eigl BJ, Finch D, Oja CD, Vergidis J, Zulfiqar M, Azad AA, Nykter M, Gleave ME, Wyatt AW, Chi KN. Circulating Tumor DNA Genomics Correlate with Resistance to Abiraterone and Enzalutamide in Prostate Cancer. Cancer Discov. 2018 Apr;8(4):444-457. doi: 10.1158/2159-8290.CD-17-0937. Epub 2018 Jan 24. PMID 29367197
- [Background] Beltran H, Wyatt AW, Chedgy EC, Donoghue A, Annala M, Warner EW, Beja K, Sigouros M, Mo F, Fazli L, Collins CC, Eastham J, Morris M, Taplin ME, Sboner A, Halabi S, Gleave ME. Impact of Therapy on Genomics and Transcriptomics in High-Risk Prostate Cancer Treated with Neoadjuvant Docetaxel and Androgen Deprivation Therapy. Clin Cancer Res. 2017 Nov 15;23(22):6802-6811. doi: 10.1158/1078-0432.CCR-17-1034. Epub 2017 Aug 25. PMID 28842510
- [Background] Khalaf DJ, Annala M, Taavitsainen S, Finch DL, Oja C, Vergidis J, Zulfiqar M, Sunderland K, Azad AA, Kollmannsberger CK, Eigl BJ, Noonan K, Wadhwa D, Attwell A, Keith B, Ellard SL, Le L, Gleave ME, Wyatt AW, Chi KN. Optimal sequencing of enzalutamide and abiraterone acetate plus prednisone in metastatic castration-resistant prostate cancer: a multicentre, randomised, open-label, phase 2, crossover trial. Lancet Oncol. 2019 Dec;20(12):1730-1739. doi: 10.1016/S1470-2045(19)30688-6. Epub 2019 Nov 11. PMID 31727538
- [Background] Khalaf D, Annala M, Finch DL, et al. Phase 2 randomized cross-over trial of abiraterone + prednisone (ABI+P) vs enzalutamide (ENZ) for patients (pts) with metastatic castration resistant prostate cancer (mCPRC): Results for 2nd-line therapy. J Clin Oncol [Internet] 2018;36(15_suppl):5015.
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Sridhar SS, Freedland SJ, Gleave ME, Higano C, Mulders P, Parker C, Sartor O, Saad F. Castration-resistant prostate cancer: from new pathophysiology to new treatment. Eur Urol. 2014 Feb;65(2):289-99. doi: 10.1016/j.eururo.2013.08.008. Epub 2013 Aug 11. PMID 23957948
- [Background] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Azad AA, Eigl BJ, Leibowitz-Amit R, Lester R, Kollmannsberger C, Murray N, Clayton R, Heng DY, Joshua AM, Chi KN. Outcomes with abiraterone acetate in metastatic castration-resistant prostate cancer patients who have poor performance status. Eur Urol. 2015 Mar;67(3):441-7. doi: 10.1016/j.eururo.2014.01.030. Epub 2014 Jan 31. PMID 24508071
- [Background] Noonan KL, North S, Bitting RL, Armstrong AJ, Ellard SL, Chi KN. Clinical activity of abiraterone acetate in patients with metastatic castration-resistant prostate cancer progressing after enzalutamide. Ann Oncol. 2013 Jul;24(7):1802-1807. doi: 10.1093/annonc/mdt138. Epub 2013 Apr 12. PMID 23585511
- [Background] Wu YM, Cieslik M, Lonigro RJ, Vats P, Reimers MA, Cao X, Ning Y, Wang L, Kunju LP, de Sarkar N, Heath EI, Chou J, Feng FY, Nelson PS, de Bono JS, Zou W, Montgomery B, Alva A; PCF/SU2C International Prostate Cancer Dream Team; Robinson DR, Chinnaiyan AM. Inactivation of CDK12 Delineates a Distinct Immunogenic Class of Advanced Prostate Cancer. Cell. 2018 Jun 14;173(7):1770-1782.e14. doi: 10.1016/j.cell.2018.04.034. PMID 29906450
- [Background] Takeda DY, Spisak S, Seo JH, Bell C, O'Connor E, Korthauer K, Ribli D, Csabai I, Solymosi N, Szallasi Z, Stillman DR, Cejas P, Qiu X, Long HW, Tisza V, Nuzzo PV, Rohanizadegan M, Pomerantz MM, Hahn WC, Freedman ML. A Somatically Acquired Enhancer of the Androgen Receptor Is a Noncoding Driver in Advanced Prostate Cancer. Cell. 2018 Jul 12;174(2):422-432.e13. doi: 10.1016/j.cell.2018.05.037. Epub 2018 Jun 14. PMID 29909987
- [Background] Viswanathan SR, Ha G, Hoff AM, Wala JA, Carrot-Zhang J, Whelan CW, Haradhvala NJ, Freeman SS, Reed SC, Rhoades J, Polak P, Cipicchio M, Wankowicz SA, Wong A, Kamath T, Zhang Z, Gydush GJ, Rotem D; PCF/SU2C International Prostate Cancer Dream Team; Love JC, Getz G, Gabriel S, Zhang CZ, Dehm SM, Nelson PS, Van Allen EM, Choudhury AD, Adalsteinsson VA, Beroukhim R, Taplin ME, Meyerson M. Structural Alterations Driving Castration-Resistant Prostate Cancer Revealed by Linked-Read Genome Sequencing. Cell. 2018 Jul 12;174(2):433-447.e19. doi: 10.1016/j.cell.2018.05.036. Epub 2018 Jun 18. PMID 29909985
- [Background] Henzler C, Li Y, Yang R, McBride T, Ho Y, Sprenger C, Liu G, Coleman I, Lakely B, Li R, Ma S, Landman SR, Kumar V, Hwang TH, Raj GV, Higano CS, Morrissey C, Nelson PS, Plymate SR, Dehm SM. Truncation and constitutive activation of the androgen receptor by diverse genomic rearrangements in prostate cancer. Nat Commun. 2016 Nov 29;7:13668. doi: 10.1038/ncomms13668. PMID 27897170
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Baca SC, Prandi D, Lawrence MS, Mosquera JM, Romanel A, Drier Y, Park K, Kitabayashi N, MacDonald TY, Ghandi M, Van Allen E, Kryukov GV, Sboner A, Theurillat JP, Soong TD, Nickerson E, Auclair D, Tewari A, Beltran H, Onofrio RC, Boysen G, Guiducci C, Barbieri CE, Cibulskis K, Sivachenko A, Carter SL, Saksena G, Voet D, Ramos AH, Winckler W, Cipicchio M, Ardlie K, Kantoff PW, Berger MF, Gabriel SB, Golub TR, Meyerson M, Lander ES, Elemento O, Getz G, Demichelis F, Rubin MA, Garraway LA. Punctuated evolution of prostate cancer genomes. Cell. 2013 Apr 25;153(3):666-77. doi: 10.1016/j.cell.2013.03.021. PMID 23622249
- [Background] Barbieri CE, Baca SC, Lawrence MS, Demichelis F, Blattner M, Theurillat JP, White TA, Stojanov P, Van Allen E, Stransky N, Nickerson E, Chae SS, Boysen G, Auclair D, Onofrio RC, Park K, Kitabayashi N, MacDonald TY, Sheikh K, Vuong T, Guiducci C, Cibulskis K, Sivachenko A, Carter SL, Saksena G, Voet D, Hussain WM, Ramos AH, Winckler W, Redman MC, Ardlie K, Tewari AK, Mosquera JM, Rupp N, Wild PJ, Moch H, Morrissey C, Nelson PS, Kantoff PW, Gabriel SB, Golub TR, Meyerson M, Lander ES, Getz G, Rubin MA, Garraway LA. Exome sequencing identifies recurrent SPOP, FOXA1 and MED12 mutations in prostate cancer. Nat Genet. 2012 May 20;44(6):685-9. doi: 10.1038/ng.2279. PMID 22610119
- [Background] Berger MF, Lawrence MS, Demichelis F, Drier Y, Cibulskis K, Sivachenko AY, Sboner A, Esgueva R, Pflueger D, Sougnez C, Onofrio R, Carter SL, Park K, Habegger L, Ambrogio L, Fennell T, Parkin M, Saksena G, Voet D, Ramos AH, Pugh TJ, Wilkinson J, Fisher S, Winckler W, Mahan S, Ardlie K, Baldwin J, Simons JW, Kitabayashi N, MacDonald TY, Kantoff PW, Chin L, Gabriel SB, Gerstein MB, Golub TR, Meyerson M, Tewari A, Lander ES, Getz G, Rubin MA, Garraway LA. The genomic complexity of primary human prostate cancer. Nature. 2011 Feb 10;470(7333):214-20. doi: 10.1038/nature09744. PMID 21307934
- [Background] Wyatt AW, Mo F, Wang K, McConeghy B, Brahmbhatt S, Jong L, Mitchell DM, Johnston RL, Haegert A, Li E, Liew J, Yeung J, Shrestha R, Lapuk AV, McPherson A, Shukin R, Bell RH, Anderson S, Bishop J, Hurtado-Coll A, Xiao H, Chinnaiyan AM, Mehra R, Lin D, Wang Y, Fazli L, Gleave ME, Volik SV, Collins CC. Heterogeneity in the inter-tumor transcriptome of high risk prostate cancer. Genome Biol. 2014 Aug 26;15(8):426. doi: 10.1186/s13059-014-0426-y. PMID 25155515
- [Background] Beltran H, Eng K, Mosquera JM, Sigaras A, Romanel A, Rennert H, Kossai M, Pauli C, Faltas B, Fontugne J, Park K, Banfelder J, Prandi D, Madhukar N, Zhang T, Padilla J, Greco N, McNary TJ, Herrscher E, Wilkes D, MacDonald TY, Xue H, Vacic V, Emde AK, Oschwald D, Tan AY, Chen Z, Collins C, Gleave ME, Wang Y, Chakravarty D, Schiffman M, Kim R, Campagne F, Robinson BD, Nanus DM, Tagawa ST, Xiang JZ, Smogorzewska A, Demichelis F, Rickman DS, Sboner A, Elemento O, Rubin MA. Whole-Exome Sequencing of Metastatic Cancer and Biomarkers of Treatment Response. JAMA Oncol. 2015 Jul;1(4):466-74. doi: 10.1001/jamaoncol.2015.1313. PMID 26181256
- [Background] Beltran H, Prandi D, Mosquera JM, Benelli M, Puca L, Cyrta J, Marotz C, Giannopoulou E, Chakravarthi BV, Varambally S, Tomlins SA, Nanus DM, Tagawa ST, Van Allen EM, Elemento O, Sboner A, Garraway LA, Rubin MA, Demichelis F. Divergent clonal evolution of castration-resistant neuroendocrine prostate cancer. Nat Med. 2016 Mar;22(3):298-305. doi: 10.1038/nm.4045. Epub 2016 Feb 8. PMID 26855148
- [Background] Gundem G, Van Loo P, Kremeyer B, Alexandrov LB, Tubio JMC, Papaemmanuil E, Brewer DS, Kallio HML, Hognas G, Annala M, Kivinummi K, Goody V, Latimer C, O'Meara S, Dawson KJ, Isaacs W, Emmert-Buck MR, Nykter M, Foster C, Kote-Jarai Z, Easton D, Whitaker HC; ICGC Prostate Group; Neal DE, Cooper CS, Eeles RA, Visakorpi T, Campbell PJ, McDermott U, Wedge DC, Bova GS. The evolutionary history of lethal metastatic prostate cancer. Nature. 2015 Apr 16;520(7547):353-357. doi: 10.1038/nature14347. Epub 2015 Apr 1. PMID 25830880
- [Background] Hong MK, Macintyre G, Wedge DC, Van Loo P, Patel K, Lunke S, Alexandrov LB, Sloggett C, Cmero M, Marass F, Tsui D, Mangiola S, Lonie A, Naeem H, Sapre N, Phal PM, Kurganovs N, Chin X, Kerger M, Warren AY, Neal D, Gnanapragasam V, Rosenfeld N, Pedersen JS, Ryan A, Haviv I, Costello AJ, Corcoran NM, Hovens CM. Tracking the origins and drivers of subclonal metastatic expansion in prostate cancer. Nat Commun. 2015 Apr 1;6:6605. doi: 10.1038/ncomms7605. PMID 25827447
- [Background] Lorente D, Omlin A, Zafeiriou Z, Nava-Rodrigues D, Perez-Lopez R, Pezaro C, Mehra N, Sheridan E, Figueiredo I, Riisnaes R, Miranda S, Crespo M, Flohr P, Mateo J, Altavilla A, Ferraldeschi R, Bianchini D, Attard G, Tunariu N, de Bono J. Castration-Resistant Prostate Cancer Tissue Acquisition From Bone Metastases for Molecular Analyses. Clin Genitourin Cancer. 2016 Dec;14(6):485-493. doi: 10.1016/j.clgc.2016.04.016. Epub 2016 May 5. PMID 27246360
- [Background] Ross RW, Halabi S, Ou SS, Rajeshkumar BR, Woda BA, Vogelzang NJ, Small EJ, Taplin ME, Kantoff PW; Cancer and Leukemia Group B. Predictors of prostate cancer tissue acquisition by an undirected core bone marrow biopsy in metastatic castration-resistant prostate cancer--a Cancer and Leukemia Group B study. Clin Cancer Res. 2005 Nov 15;11(22):8109-13. doi: 10.1158/1078-0432.CCR-05-1250. PMID 16299243
- [Background] Efstathiou E, Titus M, Wen S, Hoang A, Karlou M, Ashe R, Tu SM, Aparicio A, Troncoso P, Mohler J, Logothetis CJ. Molecular characterization of enzalutamide-treated bone metastatic castration-resistant prostate cancer. Eur Urol. 2015 Jan;67(1):53-60. doi: 10.1016/j.eururo.2014.05.005. Epub 2014 May 29. PMID 24882673
- [Background] McKay RR, Zukotynski KA, Werner L, Voznesensky O, Wu JS, Smith SE, Jiang Z, Melnick K, Yuan X, Kantoff PW, Montgomery B, Balk SP, Taplin ME. Imaging, procedural and clinical variables associated with tumor yield on bone biopsy in metastatic castration-resistant prostate cancer. Prostate Cancer Prostatic Dis. 2014 Dec;17(4):325-31. doi: 10.1038/pcan.2014.28. Epub 2014 Aug 5. PMID 25091040
- [Background] Spritzer CE, Afonso PD, Vinson EN, Turnbull JD, Morris KK, Foye A, Madden JF, Roy Choudhury K, Febbo PG, George DJ. Bone marrow biopsy: RNA isolation with expression profiling in men with metastatic castration-resistant prostate cancer--factors affecting diagnostic success. Radiology. 2013 Dec;269(3):816-23. doi: 10.1148/radiol.13121782. Epub 2013 Oct 28. PMID 23925271
- [Background] Vandekerkhove G, Chi KN, Wyatt AW. Clinical utility of emerging liquid biomarkers in advanced prostate cancer. Cancer Genet. 2018 Dec;228-229:151-158. doi: 10.1016/j.cancergen.2017.08.003. Epub 2017 Aug 25. PMID 28958406
- [Background] Carreira S, Romanel A, Goodall J, Grist E, Ferraldeschi R, Miranda S, Prandi D, Lorente D, Frenel JS, Pezaro C, Omlin A, Rodrigues DN, Flohr P, Tunariu N, S de Bono J, Demichelis F, Attard G. Tumor clone dynamics in lethal prostate cancer. Sci Transl Med. 2014 Sep 17;6(254):254ra125. doi: 10.1126/scitranslmed.3009448. PMID 25232177
- [Background] Antonarakis ES, Lu C, Wang H, Luber B, Nakazawa M, Roeser JC, Chen Y, Mohammad TA, Chen Y, Fedor HL, Lotan TL, Zheng Q, De Marzo AM, Isaacs JT, Isaacs WB, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. AR-V7 and resistance to enzalutamide and abiraterone in prostate cancer. N Engl J Med. 2014 Sep 11;371(11):1028-38. doi: 10.1056/NEJMoa1315815. Epub 2014 Sep 3. PMID 25184630
- [Background] Dijkstra S, Mulders PF, Schalken JA. Clinical use of novel urine and blood based prostate cancer biomarkers: a review. Clin Biochem. 2014 Jul;47(10-11):889-96. doi: 10.1016/j.clinbiochem.2013.10.023. Epub 2013 Oct 29. PMID 24177197
- [Background] Quek SI, Wong OM, Chen A, Borges GT, Ellis WJ, Salvanha DM, Vencio RZ, Weaver B, Ench YM, Leach RJ, Thompson IM, Liu AY. Processing of voided urine for prostate cancer RNA biomarker analysis. Prostate. 2015 Dec;75(16):1886-95. doi: 10.1002/pros.23066. Epub 2015 Aug 26. PMID 26306723
- [Background] Ulz P, Belic J, Graf R, Auer M, Lafer I, Fischereder K, Webersinke G, Pummer K, Augustin H, Pichler M, Hoefler G, Bauernhofer T, Geigl JB, Heitzer E, Speicher MR. Whole-genome plasma sequencing reveals focal amplifications as a driving force in metastatic prostate cancer. Nat Commun. 2016 Jun 22;7:12008. doi: 10.1038/ncomms12008. PMID 27328849
- [Background] Romanel A, Gasi Tandefelt D, Conteduca V, Jayaram A, Casiraghi N, Wetterskog D, Salvi S, Amadori D, Zafeiriou Z, Rescigno P, Bianchini D, Gurioli G, Casadio V, Carreira S, Goodall J, Wingate A, Ferraldeschi R, Tunariu N, Flohr P, De Giorgi U, de Bono JS, Demichelis F, Attard G. Plasma AR and abiraterone-resistant prostate cancer. Sci Transl Med. 2015 Nov 4;7(312):312re10. doi: 10.1126/scitranslmed.aac9511. PMID 26537258
- [Background] Heitzer E, Ulz P, Belic J, Gutschi S, Quehenberger F, Fischereder K, Benezeder T, Auer M, Pischler C, Mannweiler S, Pichler M, Eisner F, Haeusler M, Riethdorf S, Pantel K, Samonigg H, Hoefler G, Augustin H, Geigl JB, Speicher MR. Tumor-associated copy number changes in the circulation of patients with prostate cancer identified through whole-genome sequencing. Genome Med. 2013 Apr 5;5(4):30. doi: 10.1186/gm434. eCollection 2013. PMID 23561577
- [Background] Volik S, Alcaide M, Morin RD, Collins C. Cell-free DNA (cfDNA): Clinical Significance and Utility in Cancer Shaped By Emerging Technologies. Mol Cancer Res. 2016 Oct;14(10):898-908. doi: 10.1158/1541-7786.MCR-16-0044. Epub 2016 Jul 15. PMID 27422709
- [Background] de Bono JS, Smith MR, Saad F, Rathkopf DE, Mulders PFA, Small EJ, Shore ND, Fizazi K, De Porre P, Kheoh T, Li J, Todd MB, Ryan CJ, Flaig TW. Subsequent Chemotherapy and Treatment Patterns After Abiraterone Acetate in Patients with Metastatic Castration-resistant Prostate Cancer: Post Hoc Analysis of COU-AA-302. Eur Urol. 2017 Apr;71(4):656-664. doi: 10.1016/j.eururo.2016.06.033. Epub 2016 Jul 9. PMID 27402060
- [Background] Tran C, Ouk S, Clegg NJ, Chen Y, Watson PA, Arora V, Wongvipat J, Smith-Jones PM, Yoo D, Kwon A, Wasielewska T, Welsbie D, Chen CD, Higano CS, Beer TM, Hung DT, Scher HI, Jung ME, Sawyers CL. Development of a second-generation antiandrogen for treatment of advanced prostate cancer. Science. 2009 May 8;324(5928):787-90. doi: 10.1126/science.1168175. Epub 2009 Apr 9. PMID 19359544